CLINICAL TRIAL: NCT05677646
Title: Wearable Sensors for Delirium Detection at an Early Stage (WeSen_delirium) - an Exploratory Study
Brief Title: Wearable Sensors for Delirium Detection at an Early Stage (WeSen_delirium)
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Klinik Hirslanden, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 01
Record Dates: First submitted 2022-11-21; First posted 2023-01-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Delirium
Keywords: delirium; physical activity; sleep; activity sensor; early detection
MeSH Terms: conditions — Delirium; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delirium is an acute brain-organic syndrome: its clinical manifestation and form are results of a highly complex pathophysiology. Delirium is a serious clinical problem in hospitalized adults. It is the most common neuropsychiatric complication of hospitalization and is associated with high patient burden, increased morbidity and mortality, prolonged length of stay, higher costs, and institutionalization.

An early, accurate diagnosis as well as an adequate management are critical to the continued health and functional independence of the affected patients. Prevention strategies contain pharmacological and non-pharmacological interventions. However, their clinical success (effectiveness) is limited and the evidence for the use of pharmacological interventions for the prevention or management of delirium is scarce.

The prediction of delirium has become a new promising topic in clinical research. New approaches like the implementation of wearable sensors, in particular wearable accelerometer devices to record movements related to delirium are promising.

In this study, the study procedure only includes wearing a consumer-grade sensor on the wrist of the not-dominant hand.

This way, vital parameters are measured in order to identify patterns.

DETAILED DESCRIPTION:
Hypothesis and primary objective The overarching aim of the planned study is to identify sensor-based activity and sleep indicators and patterns (using the sensor 'Fitbit Charge 5'), which precede a delirium and thereby may qualify as potential person-level predictors to inform a predictive algorithm to detect an evolving delirium at an early stage. In addition, clarifying the feasibility of using such data for the research purpose of this study is the second aim.

Primary objectives pertain to:

1. Sensor-based profiling of delirium: Determination of delirium onset and termination; determination of sensor profiles of delirious states in terms of key characteristics (e.g., frequency of transitions between rest and inactivity, movement), which are stable across individuals whereby taking into consideration discussions on clinical motor subtypes of delirium.
2. Within-person level - forerunners and repercussions: Characterizing and comparing activity and sleep patterns (e.g., sleep deprivation, increased movement while asleep) derived from a wearable sensor preceding and following a delirium, delirium to delirium-unrelated time periods within persons who experienced a delirium (i.e., 'Can any such indicators / patterns distinguish between periods in time proximity to a delirium compared to delirium-unrelated time periods?').
3. Between-person level - forerunners and repercussions: Comparing real-time activity and sleep patterns derived from a wearable sensor across persons who experienced a delirium to those who did not (i.e., 'Can any such indicators / patterns distinguish between persons who develop a delirium and those who do not?').
4. Predictive algorithm development: Subsequently identification of activity and sleep indicators / patterns that qualify as potential forerunners of a delirium (i.e., distinct parameters or their patterns/interplay) to inform and develop a prediction algorithm for delirium detection at an early stage (to be validated in a follow-up study).
5. Visual data analysis: The investigators will employ clustering techniques (e.g., Self-Organizing Maps, K-Means Clustering) for longitudinal data to identify similar sensor measurement trajectories across study participants (e.g., for hourly heart rate measurements, hourly step counts, etc.). Because these analyses are exploratory, they will be refined on the basis of available data.

The predictions are based on a recent review summarizing state-of-the-art research. Evidence suggests the existence of clinical delirium subtypes (i.e., motor subtypes: hypoactive, hyperactive, mixed).

However, research on subtype classification is still rare. Initial research suggests that the hypoactive and mixed type seems more distinguishable from delirium than the hyperactive type. The predictions might thus be more accurate for deliria of the hypoactive and mixed type. Specifically, the investigators anticipate that:

1. Sensor-based profiling of delirium (daytime, nighttime): The investigators expect hypoactive delirious states to be characterized by decreased activity levels in comparison to non-delirium. Instead, increased activity levels during hyperactive delirious states in comparison to non-delirium are expected. Activity levels of the mixed delirium type are anticipated to range between level of the hyper- and the hypoactive type.
2. Within-person level - forerunners and repercussions (daytime):

   * Hypoactive type: The time span preceding and following a delirium during daytime will be characterized by increased activity and restlessness levels compared to delirium-unrelated time periods of an individuals during daytime.
   * Hyperactive type: The time span preceding a delirium during daytime will be characterized by increased activity and restlessness levels compared to delirium-unrelated time periods of an individuals during daytime.
3. Within-person level - forerunners and repercussions (nighttime): The time span preceding and following the delirium will be characterized by increased activity levels during nighttime (indicated by, e.g., increased mean heart rate and movement, frequency, and quantity of transitions between resting/activity), reduced sleep time / efficiency, and less minutes spent resting compared to delirium-unrelated time periods of an individual during nighttime.

However, research that carefully distinguishes time-dependent within- and between-person level predictors and their interplay through leveraging a wearable sensor is currently lacking. Also, to date, no algorithm that allows detection of deliria at an early stage has been developed. Given the novelty of this line of research, this study is mainly exploratory in nature.

Primary and secondary endpoints Endpoints Endpoints concern the sensor-based assessments (Fitbit) as well as standardized measures of delirium, such the DOS/CAM assessment (for details see Delirium-related endpoints), measured between the day of the baseline assessment and the day of discharge of the study participants.

Sensor-based endpoints:

Primary endpoints concern sensor-based in real-time indicators and their patterns related to activity and sleep assessed with the Fitbit sensor, which measures a broad range of indicators relevant to the present study, including but not limited to the example indicators listed below.

Activity- and sleep parameters, e.g.:

* heart (resting) rate, heart rate variability
* oxygen saturation, breathing rate
* skin temperature
* total sleep time, time spend in different sleep stages
* heart (resting) rate, heart rate variability
* sleep latency
* time spent in light
* 'sleep efficiency'
* step count, minutes spent in activity intensity levels (high, moderate, low)

Circadian rhythm-related indices, e.g.:

* Quantity of rest-activity transitions
* Least active 5-hours in a 24hr cycle
* Most active 10-hour period in a 24hr cycle
* Relative amplitude

Delirium-related endpoints:

Confusion Assessment Method Further endpoints concern standardized instruments for the assessment of deliria. A widely-established instrument to diagnose a delirium during an inpatient stay is the Confusion Assessment Method (CAM) which enable health care professionals to identify delirium quickly and accurately in both, clinical and research settings. The CAM is a four-point scale with the following criteria (short form): (1) acute onset and/or fluctuating course, (2) attentional disturbance, (3) formal thought disorder, (4) altered level of consciousness. All items are dichotomously scored as absent or present.

Delirium Observation Screening Scale Standard screening for delirium at the University Hospital Zurich and the Klinik Hirslanden Zurich comprises the application of a Delirium Observation Screening Scale (DOS) designed to capture early delirium symptoms, three times a day by trained nurses. If an upcoming delirium will be suspected (based on the specific DOS-value of 3 or more), it will be further assessed by CAM.

Demographic variables Non-pharmacologic factors that may influence the occurrence of delirium are increasing age, male gender, ICU or surgery interventions, transfer and changes in the setting of the patient and clinical management seems to be influenced by the subtypes of delirium.

Medical risk factors for delirium In addition, well known medical risk factors for a delirium will be collected in order to conduct a descriptive analysis. These data will be obtained from patient chart reviews of the clinical information system KISIM, namely selected variables of medical history and existing diseases of the participating patients and the medication at the time of admission, laboratory values (blood collection - clinical chemistry), and further risk-factors for delirium, e.g.: serum urea, as well as the diseases and medication at the time of discharge. The selected variables are listed in the CRF.

Sample size estimation Given the exploratory nature of the planned study, a precise sample size estimation is not possible. The aim of this study is to include 10 patients that become delirious during their USZ / Hirslanden stay as well as at least 10 patients developing no delirium during their hospital stay. Based on the data collected to date, we estimate that there is a 25% chance that new participants will develop delirium during the course of the study. Therefore, we are seeking approval to increase the maximum number of participants in the study to 72. In addition, enrollment will be stopped once we have documented 10 confirmed and analyzable cases of delirium, even if this occurs before the proposed cap of 72 participants is reached. "Analyzable" means that the participant's data are adequate for evaluation. For example, data would be considered inadequate if a participant experienced delirium but rarely or never wore the Fitbit sensor during the relevant time period.

ELIGIBILITY:
Inclusion Criteria:

* Female and male inpatients aged 65 years or older
* Cognitive ability to understand, consent to and participate in the study
* Fluent in German
* Provision of written informed consent

Exclusion Criteria:

* The presence of acute delirium,
* or a delirium diagnosis made within the last 4 weeks prior to hospitalization,
* The likelihood of an alcohol withdrawal delirium (CAGE Score >1)
* Limited knowledge of the German language
* Dementia (Mini Mental Status Test Score ≤24)

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Male and female inpatients at the Department of Internal Medicine of the University Hospital Zurich and at the Institute of General Internal Medicine Klinik Hirslanden Zurich, respectively, 65 years or older and without acute delirium or previous diagnosis of it one month prior to admission are eligible for the study.
  Patients interested in the study will be provided with the study information sheet, detailing study aims and procedure. Patients will be enrolled if they agree to participate and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
total sleep time | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
time spend in different sleep stages (deep, light, REM, awake) | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
heart rate | measured continuously over the course of the study, from enrolment to the end of the study, on average 1 week
resting heart rate | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
heart rate variability | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
oxygen saturation | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
breathing rate | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
skin temperature variation | measured daily over the course of the study, from enrolment to the end of the study, on average 1 week
Delirium Observation Scale (DOS) | measured three times per day over the course of the study, from enrolment to the end of the study, on average 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kleber, PD Dr., Principal Investigator — University of Zurich; Viktor von Wyl, Prof. Dr., Study Director — University of Zurich; Rahel Naef, Prof. Dr., Study Director — University of Zurich
Locations (2):
- Switzerland (2):
  - Klinik Hirslanden, Zurich
  - University Hospital Zurich, Internal Medicine, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davoudi A, Manini TM, Bihorac A, Rashidi P. Role of Wearable Accelerometer Devices in Delirium Studies: A Systematic Review. Crit Care Explor. 2019 Sep 13;1(9):e0027. doi: 10.1097/CCE.0000000000000027. eCollection 2019 Sep. PMID 32166280
- [Background] Godfrey A, Conway R, Leonard M, Meagher D, Olaighin GM. Motion analysis in delirium: a discrete approach in determining physical activity for the purpose of delirium motoric subtyping. Med Eng Phys. 2010 Mar;32(2):101-10. doi: 10.1016/j.medengphy.2009.10.012. Epub 2009 Nov 26. PMID 19931480
- [Background] Godfrey A, Leonard M, Donnelly S, Conroy M, Olaighin G, Meagher D. Validating a new clinical subtyping scheme for delirium with electronic motion analysis. Psychiatry Res. 2010 Jun 30;178(1):186-90. doi: 10.1016/j.psychres.2009.04.010. Epub 2010 May 10. PMID 20452050
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Marcantonio ER. Delirium in Hospitalized Older Adults. N Engl J Med. 2018 Jan 4;378(1):96-97. doi: 10.1056/NEJMc1714932. No abstract available. PMID 29298149
- [Background] Scheffer AC, van Munster BC, Schuurmans MJ, de Rooij SE. Assessing severity of delirium by the Delirium Observation Screening Scale. Int J Geriatr Psychiatry. 2011 Mar;26(3):284-91. doi: 10.1002/gps.2526. PMID 20665557
- [Background] Schuurmans MJ, Shortridge-Baggett LM, Duursma SA. The Delirium Observation Screening Scale: a screening instrument for delirium. Res Theory Nurs Pract. 2003 Spring;17(1):31-50. doi: 10.1891/rtnp.17.1.31.53169. PMID 12751884
- [Background] van Uitert M, de Jonghe A, de Gijsel S, van Someren EJ, de Rooij SE, van Munster BC. Rest-activity patterns in patients with delirium. Rejuvenation Res. 2011 Oct;14(5):483-90. doi: 10.1089/rej.2011.1181. Epub 2011 Sep 28. PMID 21954983
- [Background] Vasilevskis EE, Han JH, Hughes CG, Ely EW. Epidemiology and risk factors for delirium across hospital settings. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):277-87. doi: 10.1016/j.bpa.2012.07.003. PMID 23040281
- [Background] Zipser CM, Knoepfel S, Hayoz P, Schubert M, Ernst J, von Kanel R, Boettger S. Clinical management of delirium: The response depends on the subtypes. An observational cohort study in 602 patients. Palliat Support Care. 2020 Feb;18(1):4-11. doi: 10.1017/S1478951519000609. PMID 31506133